CLINICAL TRIAL: NCT03009526
Title: A Prospective Randomized Open-Label Study on the Efficacy and Safety of Intermittent Preventive Treatment in Pregnancy (IPTp) With Dihydroartemisinin-Piperaquine (DP) Versus IPTp With Sulfadoxine-Pyrimethamine (SP) in Malawi
Brief Title: Efficacy and Safety of IPTp-DP Versus IPTp-SP in Malawi
Acronym: STOPMIP-MW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kamuzu University of Health Sciences (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julie Gutman, Medical epidemiologist, Kamuzu University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAC-P.02/16/1872
Record Dates: First submitted 2016-12-13; First posted 2017-01-04 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Malaria; Pregnancy
Keywords: Malaria; Pregnancy; Malawi; Intermittent preventive treatment; dihydroartemisinin-piperaquine; sulfadoxine-pyrimethamine
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulfadoxine-pyrimethamine (Active Comparator): Intermittent preventive treatment with Sulfadoxine-pyrimethamine: Monthly dose of 3 co-formulated tablets containing 500 mg sulfadoxine and 25 mg pyrimethamine
  Interventions: Drug: Sulfadoxine-pyrimethamine
- dihydroartemisinin-piperaquine (Experimental): Intermittent preventive treatment with dihydroartemisinin-piperaquine: Monthly course of daily doses of co-formulated DP tablets containing 40 mg dihydroartemisinin and 320 mg piperaquine, dosed based on the woman's weight, for 3 days:
  * 24-35.9 kg: Two tablets
  * 36-59.9 kg: Three tablets
  * 60-79.9 kg: Four tablets
  * ≥80 kg: Five tablets
  Interventions: Drug: dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine — 500 mg sulfadoxine and 25 mg pyrimethamine
  Other Names: Fansidar
  Arms: Sulfadoxine-pyrimethamine
Drug: dihydroartemisinin-piperaquine — 40 mg dihydroartemisinin and 320 mg piperaquine
  Arms: dihydroartemisinin-piperaquine

SUMMARY:
This study aims to compare the efficacy of monthly IPTp-DP with monthly IPTp-SP to determine if IPTp-DP is associated with a reduction in malaria infection at delivery among HIV-negative women in an area with high levels of SP resistance in Malawi.

DETAILED DESCRIPTION:
Problem to be studied Malaria in pregnancy (MiP) due to Plasmodium falciparum infection is a major cause of maternal morbidity and poor birth outcomes in malaria-endemic countries. Pregnant women are at increased risk of more frequent and severe malaria infections than non-pregnant women. Intermittent preventive treatment in pregnancy (IPTp) with sulfadoxine-pyrimethamine (SP), which involves administration of treatment doses of SP at each antenatal visit in the second and third trimesters of pregnancy, at least one month apart, irrespective of malaria parasitemia, is currently recommended for all women, except HIV positive women taking daily cotrimoxazole prophylaxis, in areas with stable moderate to high transmission of malaria.

SP is the only drug currently used for IPTp. Due to increasing resistance to SP, it is no longer used as a treatment for symptomatic malaria, however, IPTp-SP remains effective even in areas where SP resistance in children under five (determined by in vivo efficacy studies) is up to 26%, and continues to be used for IPTp in countries where SP is no longer recommended to treat symptomatic malaria. However, IPTp-SP has become more controversial given recent data from northern Tanzania and Malawi that have demonstrated that at higher rates of resistance, IPTp-SP may no longer be effective.

Alternative drugs which could replace SP have been tested; mefloquine, azithromycin-chloroquine, and amodiaquine have been abandoned as options due to poor tolerability among pregnant women. Dihydroartemisinin-Piperaquine (DP) remains an attractive option because of the long half-life of piperaquine (PQ) and the demonstrated efficacy, safety, and tolerability in pregnancy. Recent studies in Kenya and Uganda using DP for IPTp demonstrated a significant reduction in the prevalence of malaria throughout pregnancy and at the time of delivery. However, there was not a clear benefit in terms of improved neonatal outcomes. Additional studies are therefore needed to determine the impact of switching from IPTp-SP to IPTp-DP.

Study aims Primary objectives To compare the efficacy of monthly IPTp-DP with monthly IPTp-SP to determine if IPTp-DP is associated with a reduction in malaria infection at delivery among HIV-negative women in an area with high levels of SP resistance in Malawi.

Secondary objectives

* To determine if IPTp-DP results in decreased fetal morbidity compared with IPTp-SP, where fetal morbidity is defined as the composite of any of the following: Preterm birth (< 37 weeks gestation), low birth weight (LBW) (< 2,500 grams), or small for gestational age (SGA).
* To evaluate the tolerability and safety of IPTp-DP in the second and third trimesters of pregnancy, including an assessment of cardiac risk, as measured by changes in QTc intervals from baseline with each successive dose.
* To compare the frequency of adverse events and fetal congenital malformations in IPTp-DP with IPTp-SP.
* To assess how SP and DP affect the maternal intestinal and vaginal microbiome.

Methodology Open-label, 2 arm randomized controlled superiority trial to compare the efficacy and safety of IPTp-DP to IPTp-SP in Malawi. The trial is designed to show a 60% decrease in malaria infection at delivery among HIV-negative women of all gravidity when IPTp-DP is used instead of IPTp-SP.

Expected findings and dissemination It is expected that in areas of high SP resistance, IPTp-DP will be superior to IPTp-SP in decreasing malaria infection at delivery. In addition, it is anticipated that DP will be well-tolerated among pregnant women and that fetal outcomes will be better than IPTp-SP.

ELIGIBILITY:
Inclusion Criteria:

* Viable singleton pregnancy
* Gestational age ≤28 completed weeks (28 6/7) by fundal height/ultrasound
* Maternal age ≥16 years
* No history of IPTp use during this pregnancy
* Willing to participate and complete the study schedule, including laboratory studies and delivery in the labor ward of the study clinic or hospital
* Willing to sign or thumb print informed consent
* Resident of study area and intending to stay in the area for the duration of the follow-up
* HIV-negative at enrolment

Exclusion Criteria:

* HIV-positive or unknown
* Multiple gestation
* High-risk pregnancy, including any pre-existing illness likely to cause complication of pregnancy (hypertension, diabetes, asthma, epilepsy, renal disease, liver disease, fistula repair, leg or spine deformity)
* Severe anemia requiring blood transfusion (Hb <7.0 g/dL) at enrolment
* Known allergy or previous adverse reaction to any of the study drugs
* Previous inclusion in the same study
* Participating in other malaria intervention studies
* Known or suspected cardiac disease
* Corrected QT interval (QTcF) greater than 450 ms at baseline
* Patients taking any of the following drugs:

  * Antimicrobial agents of the following classes (systemic use only):

    * Macrolides (e.g. erythromycin, clarithromycin, azithromycin, roxithromycin)
    * Fluoroquinolones (e.g., levofloxacin, moxifloxacin, sparfloxacin)
    * Pentamidine
  * Antiarrhythmic agents (e.g. amiodarone, sotalol)
  * Antihistamines (e.g. promethazine)
  * Antifungals (systemic): ketoconazole, fluconazole, itraconazole
  * Antiretrovirals: Saquinavir
  * Diuretics (e.g. hydrochlorothiazide, furosemide)
  * Antipsychotics (neuroleptics): haloperidol, thioridazine
  * Antidepressants: imipramine, citalopram, escitalopram
  * Antiemetics: domperidone, chlorpromazine, ondansetron

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Malaria infection at the time of delivery | delivery
  The composite of peripheral and placental parasitemia, detected by placental histology, positive peripheral blood smear at the time of delivery, or positive rapid diagnostic test at the time of delivery
Fetal morbidity | Delivery
  Composite endpoint of fetal morbidity, defined as any of the following: Preterm birth (birth before 37 weeks gestation), Low-birth-weight (birth weight under 2,500 grams), Small for gestational age (SGA)

SECONDARY OUTCOMES:
Electrocardiogram changes following the receipt of DP | 4-6 hours after the 3rd dose with each course
  QTc will be measured in a subset of women 4-6 hours after the 3rd dose of each course
Microbiome changes following receipt of DP or SP | From date of randomization until the date of delivery or last date of follow-up, average of ~4-5 months
  We will measure the changes in the intestinal and vaginal microbiome induced by DP and SP
Maternal hemoglobin at 3rd trimester | 3rd trimester
Maternal anemia at 3rd trimester | 3rd trimester
Fetal anemia | Delivery
  Anemia/ hemoglobin measured from cord blood
Incidence of clinical malaria episodes | From date of randomization until the date of delivery or last date of follow-up, average of ~4-5 months
Incidence of all cause sick visits | From date of randomization until the date of delivery or last date of follow-up, average of ~4-5 months
Serious adverse events | From date of randomization until the date of delivery or last date of follow-up, average of ~4-5 months

CONTACTS AND LOCATIONS:
Overall Officials: Don P Mathanga, MBBS PhD, Principal Investigator — Malawi College of Medicine; Julie Gutman, MD MSc, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Malaria Alert Center, University of Malawi College of Medicine, Liwonde, Malawi

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researches upon submission and approval of a detailed request
Supporting Information: Study Protocol, SAP
Time Frame: January 2022
Access Criteria: IPD will be shared with other researches upon submission and approval of a detailed request

REFERENCES:
- [Derived] Andronescu LR, Sharma A, Peterson I, Kachingwe M, Kachepa W, Liang Y, Gutman JR, Mathanga DP, Chinkhumba J, Laufer MK. The Effect of Intermittent Preventive Treatment of Malaria During Pregnancy and Placental Malaria on Infant Risk of Malaria. J Infect Dis. 2022 Jan 18;225(2):248-256. doi: 10.1093/infdis/jiab351. PMID 34216212